CLINICAL TRIAL: NCT02449512
Title: Somatosensory Evoked Potentials From the Lower Urinary Tract in Individuals With Neurogenic Lower Urinary Tract Dysfunction as a Result of Spinal Cord Injury
Brief Title: Somatosensory Evoked Potentials From the Lower Urinary Tract
Status: Withdrawn | Type: Observational
Why Stopped: Funding issues
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2014-20
Record Dates: First submitted 2015-05-15; First posted 2015-05-20 (Estimated); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Neurogenic Lower Urinary Tract Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- complete: individuals with somato-sensory complete spinal cord injury
- incomplete: individuals with somato-sensory incomplete spinal cord injury

SUMMARY:
Spinal cord injury and other systemic neurological diseases (Multiple Sclerosis, Parkinson's disease) affect the integrity of lower urinary tract (LUT) function, leading to neurogenic lower urinary tract dysfunction (NLUTD). The urodynamic investigation is the current "gold-standard" for evaluating LUT function. Nevertheless, the sensory situation of the LUT cannot be investigated objectively. Furthermore, the current classification of the severity of the NLUTD due to spinal cord injury (SCI) does not represent the sensory situation of the LUT. Additional investigations therefore need to be established for assessing the sensory situation of the LUT. Somatosensory evoked potentials (SEPs) are an established method for investigating the processing of sensory nervous activity. However, SEPs from the LUT of SCI individuals have not yet been investigated.

A novel technique, i.e. diffusion tensor imaging (DTI), allows to process magnetic resonance images (MRI) in order to visualize nerve fibers. Using DTI, the innervation of the bladder after SCI can be visualized. The structural presentation of bladder innervation will be compared with the functional results, i.e. the SEP of the LUT in SCI individuals.

The primary objective of the proposed study is to elicit and characterize (latency, amplitude) the somatosensory evoked potentials (SEPs) from the bladder in individuals suffering from neurogenic lower urinary tract dysfunction as a result of spinal cord injury.

Furthermore, the SEPs from the bladder will be compared with the SEPs from peripheral nerves (N. tibialis, N. pudendus, N. medianus).

Moreover, the latency and amplitude of the SEPs from the bladder of individuals with somato-sensory complete spinal cord injury will be compared with those from the bladder of individuals with somato-sensory incomplete spinal cord injury.

Finally, the structural innervation of the bladder after SCI will be compared with the remaining sensory function.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Chronic SCI of a minimum of 1 year
* Aetiology of SCI: traumatic

Exclusion Criteria:

* Age < 18 years or > 70 years
* Aetiology of SCI: non-traumatic
* History of bleeding disorder
* History of chronic neuropathic pain
* Intravesical botulinum toxin injections < 12 months ago
* Bladder management using indwelling catheters (suprapubic, transurethral)
* Bladder augmentation
* Sacral deafferentation
* Sacral neuromodulation
* Acute, symptomatic urinary tract infection
* Pregnancy
* Urolithiasis
* Bladder cancer
* Exclusion criteria for MRI (cardiac pace maker, implanted metal etc.)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individuals with neurogenic lower urinary tract dysfunction as a result of spinal cord injury
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
occurrence of somatosensory evoked potentials from the bladder | within 1 week after enrollment into study

SECONDARY OUTCOMES:
latency of somatosensory evoked potentials | within 1 week after enrollment into study
peak-to-peak amplitude of somatosensory evoked potentials | within 1 week after enrollment into study
nerve fiber density around bladder | within 1 week after enrollment into study
fractional anisotropy of nerve fibers around bladder | within 1 week after enrollment into study
apparent diffusion coefficient of nerve fibers around bladder | within 1 week after enrollment into study

OTHER OUTCOMES:
age | 1st day
gender | 1st day
severity of spinal cord injury | 1st day
  American Association of Spinal Cord Injury Impairment Score

CONTACTS AND LOCATIONS:
Overall Officials: Jens Wöllner, Principal Investigator — Swiss Paraplegic Centre
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No